CLINICAL TRIAL: NCT02540057
Title: Flexor Carpi Radialis or Abductor Pollicis Longus in Ligament Reconstruction and Tendon Interposition - A Randomized Controlled Trial
Brief Title: FCR or APL in LRTI - A Single Surgeon Randomized Controlled Trial
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Abandoned following local ethics review.
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Principal Investigator, David Tang, MD, Nova Scotia Health Authority
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FCRAPLRCT
Record Dates: First submitted 2015-09-01; First posted 2015-09-03 (Estimated); Last update posted 2016-08-05 (Estimated); Status verified 2016-08

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Flexor carpi radialis (Active Comparator): These patients will have their trapeziectomy with ligament reconstruction and tendon interposition using the flexor carpi radialis tendon.
  Interventions: Procedure: Flexor carpi radialis
- Abductor pollicis longus (Active Comparator): These patients will have their trapeziectomy with ligament reconstruction and tendon interposition using the abductor pollicis longus tendon.
  Interventions: Procedure: Abductor pollicis longus

INTERVENTIONS:
Procedure: Flexor carpi radialis — Ligament reconstruction with tendon interposition completed using the flexor carpi radialis tendon
  Arms: Flexor carpi radialis
Procedure: Abductor pollicis longus — Ligament reconstruction with tendon interposition completed using the abductor pollicis longus tendon
  Arms: Abductor pollicis longus

SUMMARY:
We are investigating the use of the flexor carpi radialis and abductor pollicis longus tendons in the use of trapeziectomy and ligament reconstruction with tendon interposition. Previous studies have shown clinical equipoise, and we plan to do a randomized controlled trial to further assess.

DETAILED DESCRIPTION:
Trapeziometacarpal osteoarthritis (TMC OA) is a great societal burden. Its prevalence has been reported as high as 36% in select populations, and is directly responsible for reduced work productivity and absenteeism in many cases. In 1949 Gervis originally described simply removing the offending bone, the trapezium, and trapeziectomy has since shown favorable outcomes. Many others have subsequently published similar clinical results with the same technique. However, it has been noted that with trapeziectomy alone there is the risk of metacarpal subsidence into the trapezial fossa over time, which may have an impact on patient outcomes. This observation was the impetus for the development of several more complex surgical interventions for TMC OA.

A recent Cochrane review investigated the literature available comparing seven surgical interventions for TMC OA. There were very few significant differences discovered, and they ultimately did not identify a single procedure as superior. The included studies however were noted as being of low quality, and the authors called for more robust trials with standardized outcome measures.

One of the more popular techniques reviewed is the trapeziectomy with ligament reconstruction and tendon interposition (LRTI). First described by Eaton and Littler, it has been met with widespread adoption, and has shown good results. It theoretically reconstructs the ligament responsible for maintaining the metacarpal's position, and also places a tendon interposed between the two bones (scaphoid and base of the first metacarpal) thus limiting its collapse. The most commonly used tendon for reconstruction of the volar beak ligament is the flexor carpi radialis (FCR), but recent reports have also advocated for use of the abductor pollicis longus (APL). The APL tendon already inserts onto the base of the first metacarpal, obviating the need for creating a bone tunnel, which is required when using the FCR. It can also be harvested without the need for additional incisions. Only one study has directly compared the two procedures, and the results were similar for both.

Based on the available literature, trapeziectomy with LRTI may confer minor advantages to simple trapeziectomy. Currently, surgeons at our institution unanimously prefer the LRTI procedure, however there is discord on which tendon is best suited for the reconstruction. We hypothesize that complications will be similar between the two procedures, but DASH scores and operative time will be significantly decreased when using the APL tendon for reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* patients with any grade of trapeziometacarpal joint osteoarthritis undergoing surgical correction with trapeziectomy and ligament reconstruction with tendon interposition

Exclusion Criteria:

* previous wrist surgery, inflammatory arthritis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-08; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Disabilities of arm shoulder and hand questionnaire | 5 years
  questionnaire

SECONDARY OUTCOMES:
thumb range of motion | 5 years
grip strength | 5 years
  jamar dynamometer

CONTACTS AND LOCATIONS:
Overall Officials: Joseph P Corkum, MD,BEng, Study Director — Nova Scotia Health Authority

REFERENCES:
- [Background] Vermeulen GM, Spekreijse KR, Slijper H, Feitz R, Hovius SE, Selles RW. Comparison of arthroplasties with or without bone tunnel creation for thumb basal joint arthritis: a randomized controlled trial. J Hand Surg Am. 2014 Sep;39(9):1692-8. doi: 10.1016/j.jhsa.2014.04.044. Epub 2014 Jun 10. PMID 24928359
- [Result] Wajon A, Vinycomb T, Carr E, Edmunds I, Ada L. Surgery for thumb (trapeziometacarpal joint) osteoarthritis. Cochrane Database Syst Rev. 2015 Feb 23;2015(2):CD004631. doi: 10.1002/14651858.CD004631.pub4. PMID 25702783